CLINICAL TRIAL: NCT02117973
Title: iAssist vs. Conventional Instrumentation in Total Knee Arthroplasty Using the Persona Knee System Among Patients With BMI>=30: Radiographic, Clinical and Economic Outcomes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0092-13-HMO
Record Dates: First submitted 2014-02-26; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-02

CONDITIONS: Primary Knee Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Technique using Persona prosthesis (Active Comparator): The surgeon will realize the implantation of the Persona prosthesis according to the surgical technique. Potential variables such as methodology for determining tibial rotation, measuring of bone cuts, and any intra-operative adjustments will be captured on the operative case report form.
  Interventions: Procedure: iAssist Technique using Persona system vs. the conventional technique using Persona system
- iAssist Technique using Persona prosthesis (Experimental): iAssist is an electronic displacement sensor based instrumentation system that provides intra-operative verification at each surgical step (bone cuts alignment and resection level); in order to help reduce bone cuts errors. iAssist features simple and intuitive instrumentation that is based on conventional total knee arthroplasty instrumentation. iAssist should take less than 2-3 minutes (on average) to setup
  Interventions: Procedure: iAssist Technique using Persona system vs. the conventional technique using Persona system

INTERVENTIONS:
Procedure: iAssist Technique using Persona system vs. the conventional technique using Persona system

SUMMARY:
The purpose of this prospective randomized study is to evaluate iAssist with respect to radiographic, clinical and economic outcomes in comparison to conventional instrumentation in primary total knee arthroplasty using the Persona knee system among patients with BMI>=30.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Needs a primary TKR on the left or right knee
3. Diagnose of non-inflammatory degenerative joint disease (e.g., osteoarthritis, post-traumatic arthritis, avascular necrosis, etc.)
4. Over 18 years old
5. BMI>=30
6. Able to:

   * Understand what participation in the study entails and give written informed consent, and
   * Follow surgeon/staff instructions, and
   * Return for all follow-up evaluations, and
   * Able and willing to undergo a preoperative full-leg, standing radiographs (all cases)
   * Willing to consent (patient or his/her legal guardian) to participate in the study by signing and dating an approved consent.
   * Meet an acceptable preoperative medical clearance and is free of or treated for cardiac, pulmonary, hematological or other conditions that would pose excessive operative risk.
7. Presence of varus or valgus deformity of 15 degrees or less.

Exclusion Criteria:

1. Currently enrolled in an investigational new drug or device study
2. Active Infection (including septic knee, distant infection, or osteomyelitis)
3. Severe hip arthrosis
4. Neurological disorders (including, but not limited to Parkinson's disease)
5. Prior ipsilateral unicompartmental knee arthroplasty, TKA, knee fusion or patellectomy
6. Hip or knee ankylosis
7. Inflammatory joint disease.
8. Either rheumatoid or post-traumatic knee arthritis
9. Scheduled for simultaneous bilateral TKA
10. Indications of intra- and/or extra-articular deformations that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately sized implant, such as polio, history of tibial plateau fracture, etc.
11. Any metal within 150 mm of the joint line for the operative-side knee
12. Knee deformities greater than 15 degrees of fixed varus, valgus, or flexion contracture on initial physical examination
13. A female who is pregnant or lactating
14. Current involvement in any personal injury litigation, medical-legal or worker's compensation claims
15. Arterial disease or stents that would exclude the use of a tourniquet
16. Insufficient quality or quantity of bone to support the implant due to prior knee surgery (or surgeries), cancer, metabolic bone disease, osteoporosis/osteopenia (diagnosed or treated with medication), active/old/remote infection, etc.
17. Mental condition that may interfere with his/her ability to give an informed consent or interfere with his/her ability or willingness to fulfill the requirements of the study.
18. Condition that would place excessive demands on the implant (e.g., Charcot's joints, muscle deficiencies, multiple joint disabilities, skeletal immaturity, etc.).
19. Collateral ligament insufficiency.
20. Immunosuppressive disorder (e.g., AIDS, etc.) that would require cytotoxic drugs, corticosteroids, large dose of irradiation, or antilymphocytic serum.
21. An existing condition that would, in the opinion of the investigator, compromise participation or follow-up in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
differences in limb alignment | 12 MONTHS
  The primary endpoint is defined as Limb alignment as determined using radiographs (A/P long-standing and lateral films)

SECONDARY OUTCOMES:
difference in Knee Society Score | 12 MONTHS
  Assess the differences in Knee Society Score between iAssist and conventional instrumentation in primary TKA procedures.

OTHER OUTCOMES:
difference in Oxford knee score | 12 months
  Assess the differences inOxford knee score between iAssist and conventional instrumentation in primary TKA procedures.
Operating room time | three hours
  to compare the operating room time between patients undergoing iAssist vs. conventional instrumentation in primary TKA procedures.
Blood loss and complications | 12 months
  to compare the blood loss and complications between patients undergoing iAssist vs. conventional instrumentation in primary TKA procedures